CLINICAL TRIAL: NCT01551901
Title: LIFT: Luna Interbody System for Fusion Trial
Brief Title: Luna Interbody System for Fusion Trial
Acronym: LIFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Benvenue Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEN 007
Record Dates: First submitted 2012-02-02; First posted 2012-03-13 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Lower Back Pain; Degenerative Disc Disease (DDD)
Keywords: Back pain; Spinal fusion; Degenerative disc disease (DDD); Lower back pain; Fusion
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Degeneration; Back Pain | interventions — Spinal Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Luna Interbody System (Experimental)
  Interventions: Device: Spinal fusion

INTERVENTIONS:
Device: Spinal fusion — Spinal fusion procedures in skeletally mature patients with symptomatic degenerative disc disease (DDD) at one or two contiguous levels from L2-S1 with up to grade 1 spondylolisthesis
  Other Names: Luna Interbody System

SUMMARY:
The purpose of this trial is to evaluate the performance, safety and effectiveness of the Luna system for the treatment of degenerative disc disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 65 at the time of consent
2. Patient has back pain consistent with symptomatic degenerative disc disease at one level or two contiguous levels from L2-S1 requiring surgical intervention.
3. Patient has had at least 6 months of non-operative care
4. Patient is mentally capable and willing to sign a study-specific informed consent form
5. Patient is willing and able to comply with all study requirements
6. Patient has a score on the back pain visual analog scale (VAS) of ≥ 40 mm
7. Patient has an Oswestry Disability Index (ODI) score of ≥ 30%

Exclusion Criteria:

1. DDD affecting >2 levels
2. Back pain due to causes other than DDD
3. Spine surgery within last 3 months or planned spine surgery within 6 weeks of post study procedure
4. >Grade 1 spondylolisthesis or retrolisthesis
5. Infection at or close to target disc level
6. Active systemic infection
7. Patient has known osteoporosis
8. Prior interbody fusion at the target level
9. Prior failed interbody fusion at any level
10. Known allergy to device materials
11. Uncontrolled psychiatric illness or severe dementia
12. Pregnant at time of enrollment or considering getting pregnant during study period
13. Any metabolic or other bone disease that could significantly compromise pedicle screw and/or interbody device placement.
14. Any severe illness that would prevent complete study participation
15. Uncontrolled diabetes
16. Current use of chronic steroids (more than equivalent of 10 mg prednisone daily)
17. Contraindication to spinal surgery or general anesthesia
18. Coagulopathy
19. Body mass index >35
20. Current smoker
21. Known illicit substance abuser
22. Currently participating in another investigational study that could affect responses to the study device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with device in place showing lack of device migration or subsidence and absence of device related serious adverse event | 12 Month Post-op
Improvement in pain score on the Visual Analog Scale (VAS) from baseline | 12 Month Post-op
Maintenance or improvement of neurologic function related to the spine | 12 Month Post-op
Proportion of subjects with lack of revision, removal, reoperation or use of additional supplemental fixation | 12 Month Post-op
Improvement in Oswestry Disability Index (ODI) score from baseline | 12 Month Post-op

SECONDARY OUTCOMES:
Improvement from baseline in quality of life as measured by SF-36 | 12 Month Post-op
Rate of device-related serious adverse events | 12 Month Post-op
Proportion of subjects with radiographic fusion of target segments | 12 Month Post-op

CONTACTS AND LOCATIONS:
Overall Officials: Alphonse Lubansu, M.D., Principal Investigator — Erasme University Hospital
Locations (5):
- Belgium (3):
  - Clinique du Parc Leopold, Brussels
  - Hôpital Erasme, Brussels
  - CHC Liege, Liège
- Germany (2):
  - Universitatsklinikum Bonn, Bonn
  - Paracelsus Kliniken, Zwickau